CLINICAL TRIAL: NCT07183124
Title: Using 3D Modeling to Detect Locally Advanced Rectal Cancer With Positive Circumferential Resection Margin
Brief Title: 3D Modeling for Detecting Locally Advanced Rectal Cancer With Positive Circumferential Resection Margin
Status: Not yet recruiting | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Other Study IDs: CE25536A; TCVGH-NHRI1142008 (Other Grant/Funding Number: Taichung Veterans General Hospital)
Record Dates: First submitted 2025-09-14; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: General Surgery; Oncology; Medical Informatics
Keywords: rectal cancer; 3D Modeling; deep learning; Pelvic CT Imaging; Clinical Prediction Model
MeSH Terms: conditions — Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: AI-Assisted 3D Imaging Model for Tumor and CRM Assessmen — This study uses an AI-assisted 3D imaging model to analyze existing CT and MRI images of stage II-III locally advanced rectal cancer patients. The system reconstructs tumor boundaries and spatial relationships, predicts circumferential resection margin (CRM) status, and supports staging assessment. No interventions are performed on participants, and all data are collected retrospectively from routine clinical care.

SUMMARY:
This retrospective study aims to develop an AI-assisted 3D modeling system to improve staging accuracy for stage II-III locally advanced rectal cancer (LARC). High-quality CT images from Taichung Veterans General Hospital will be used to reconstruct tumor boundaries and spatial relationships. The AI model will be trained and validated against MRI and pathology results to predict circumferential resection margin (CRM) status. Outcomes include sensitivity, specificity, accuracy, and agreement with standard imaging. This system seeks to support precise tumor staging and inform future clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with rectal cancer, clinical stage II-III, with no distant metastasis (M0)
* Age over 18 years, with adequate physical status classified as American Society of Anesthesiologists (ASA) I-III, capable of receiving treatment and surgery
* No history of other malignancies or major diseases affecting study assessment within the past three years.
* Complete medical records, including available CT and MRI imaging.

Exclusion Criteria:

* Patients with clinical stage I or IV rectal cancer.
* Age under 18 years, or physical status not meeting American Society of Anesthesiologists (ASA) I-III criteria, unable to undergo surgery or related treatment.
* Presence of other major diseases or malignancies affecting tumor assessment (e.g., diagnosis of another malignancy within the past three years, uncontrolled cardiovascular disease).
* Incomplete medical records or imaging data, including missing required CT or MRI images.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients (≥18 years) diagnosed with stage II-III locally advanced rectal cancer (LARC) without distant metastasis (M0), who received care at Taichung Veterans General Hospital (TVGH), Taiwan. Eligible participants have adequate physical status (ASA I-III) to undergo standard treatment and surgery, no history of other malignancies or major diseases affecting tumor assessment within the past three years, and complete medical records including CT and MRI imaging. Patients with stage I or IV disease, insufficient physical status, major comorbidities, or incomplete imaging/medical records are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of the AI-assisted 3D imaging model for predicting circumferential resection margin (CRM) negativity | Day 1 (At the time of retrospective imaging analysis)
  Model predictions are compared with pathology results (gold standard) to assess diagnostic accuracy.

SECONDARY OUTCOMES:
Accuracy and agreement of AI model predictions with MRI interpretations | Day 1 (At the time of retrospective imaging analysis)
  Agreement between AI model, MRI, and pathology results will be analyzed using Kappa statistics to evaluate consistency and reliability.

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan